CLINICAL TRIAL: NCT06401343
Title: Sodium-dependent Glucose Transporters 2 Inhibitor in Nonobstructive Hypertrophic Cardiomyoapthy Patients With Heart Failure With Preserved Ejection Fraction: a Prospective, Multi-center,Open-lable,Randomized Controlled Trial
Brief Title: Use of SGLT2i in noHCM With HFpEF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Lianming Kang, Dr. Lianming Kang, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-ZX006
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Hypertrophic Cardiomyopathy; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Use of Empagliflozin+guideline directed medical treatment of HCM
  Interventions: Drug: Empagliflozin 10 MG
- Control group (No Intervention): Guideline directed medical treatment of HCM

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Participants randomized to the study group will received Empagliflozin 10mg q.d. for 12 months.
  Arms: Study group

SUMMARY:
This study aims to evaluate the impact of Sodium-dependent glucose transporters 2 inhibitor Empagliflozin on the exercise capacity,symptoms of heart failure, cardiac function, myocardial remodeling and quality of life of nonobstructive HCM patients with HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of nonobstructive hypertrophic cardiomyopathy;
* At least 18 years old;
* LVEF≥50%
* Elevated NT-proBNP >300 pg/ml for patients without atrial fibrillation (AF), or >900 pg/ml for patients with AF at Visit 1;
* NYHA II-IV
* Capable of performing cardiopulmonary exercise test with an RER≥1.0
* Signed and dated written informed consent and willing to return for clinical follow-up.

Exclusion Criteria:

* Under-went septal reduction therapy within 3 months before screening;
* Acute decompensation heart failure within 3 months before screening;
* Symptomatic low BP or SBP<100mmHg;
* eGFR<30ml/min/1.73m2
* LVOTG ≥30mmHg at rest or under provocation;
* Renal insufficiency with eGFR<50mL/min/1.73m2
* ICD implantation or CRT planned within 3 months;
* Women who are pregnant, or who plan to become pregnant while in the trial;
* Currently enrolled in another investigational device or drug trial;
* Combining any other clinical condition with a life expectancy less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
VO2max on cardiopulmonary exercise tesing | 12 months

SECONDARY OUTCOMES:
NT-ProBNP | 12 months
NYHA heart failure classification | 12 months
KCCQ-CSS | 12 months
HCMSQ-(SoB) | 12 months
E/A | 12 months
E/e' | 12 months
Peak tricuspid regurgitation velocity | 12 months
Left atrium volume index , LAVI | 12 months
Left Ventricular Mass index, LVMI | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Centre for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No